CLINICAL TRIAL: NCT06485570
Title: Knowledge of Nursing Theories of Teaching With Creative Drama in Fundamentals of Nursing Course Level and Perception of Nursing Profession
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Ebru Sevinç, Lecturer, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Istanbul Arel University
Record Dates: First submitted 2024-04-02; First posted 2024-07-03 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Explaining Nursing Theories Through Creative Drama
Keywords: creative drama nursing theories perception of nursing

STUDY DESIGN:
Intervention Model Description: 50 first year nursing students, 25 experimental, 25 control
Who Masked: Participant
Masking Description: 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): In the control group, the trainings prepared by the researcher in line with the literature information on the Environmental Theory, Self-Care Disability Theory and Adaptation Model will be carried out in 3 sessions with the lecture method, respectively. The trainings will be planned in the classroom environment for 4 weeks and 2 lesson hours (100 minutes) for each session. At the end of the trainings, "Knowledge Measurement Questionnaire" and "Perception of Nursing Profession Scale" will be applied to the participants as a post-test to measure their level of knowledge about nursing theories. In the third stage of the study, semi-structured interviews will be conducted with the students from the experimental group after the applications in order to reveal the participants' views on teaching methods.
  Interventions: Other: control
- Experimental (Experimental): The trainings prepared by the researcher in line with the literature information on Environmental Theory, Self-Care Disability Theory and Adaptation Model will be carried out in 3 sessions with creative drama teaching method to the experimental group. The trainings will be planned in the classroom environment for 4 weeks and 2 lesson hours (100 minutes) for each session. At the end of the trainings, "Knowledge Measurement Questionnaire" and "Perception of Nursing Profession Scale" will be applied to the participants as a post-test to measure their level of knowledge about nursing theories. In the third stage of the study, semi-structured interviews will be conducted with the students from the experimental group after the applications in order to reveal the participants' views on teaching methods.
  Interventions: Other: creative drama training

INTERVENTIONS:
Other: creative drama training — The trainings prepared by the researcher in line with the literature information on Environmental Theory, Self-Care Disability Theory and Adaptation Model will be carried out in 3 sessions with creative drama teaching method to the experimental group. The trainings will be planned in the classroom environment for 4 weeks and 2 lesson hours (100 minutes) for each session. At the end of the trainings, "Knowledge Measurement Questionnaire" and "Perception of Nursing Profession Scale" will be applied to the participants as a post-test to measure their level of knowledge about nursing theories. In the third stage of the study, semi-structured interviews will be conducted with the students from the experimental group after the applications in order to reveal the participants' views on teaching methods.
  Arms: Experimental
Other: control — control group
  Arms: control group

SUMMARY:
The aim of the study was to teach nursing students nursing theories through creative drama method. The aim of the study was to investigate the effect of the teaching on the level of knowledge and perception of nursing profession. In the research A mixed research method using both quantitative and qualitative methods will be used. The quantitative dimension of the research will be a randomized controlled experimental (pre-test-post-test control group design) is a study. The qualitative dimension is based on the individual interviews with the experimental and control groups. will constitute the interview method.

In the study, it is planned to use the "Knowledge Measurement Questionnaire" prepared by the researcher in line with the literature, the "Perception of Nursing Profession Scale" developed by Eşer et al. (2006), and the "Personal Information Form" containing descriptive information as data collection forms.

Data Analysis of Expert Opinion: The draft drama training program prepared by the trainer related to the Adaptation Model, Environmental Theory, Self-Care Disability Theory will be presented for expert opinion. In addition, the draft achievement test created in line with the literature will be presented to 10 experts and the content validity will be analyzed with the Davis Technique.SSPS 22.0 package program in scale analysis will be used. Skewness and Kurtosis (kurtosis, skewness), normal distribution curve and Levene's test values.

Qualitative Data Analysis: Content analysis will be conducted using MAXQDA program.

50 students who voluntarily accepted to participate in line with the inclusion and exclusion criteria will be invited to the study. In the first stage of the study, 50 students will be asked to fill in the "Personal Information Form", "Knowledge Measurement Questionnaire" and "Perception of Nursing Profession Scale" before any training on the subject and they will be informed about the definition and importance of nursing models/theories. training will be conducted. Then, the students participating in the study will be randomized to the experiment (n:25) and control (n:25) groups. In the second phase of the research, the experiment group with creative drama method and the control group with traditional teaching method. using respectively; Environmental Theory, Self-Care Disability Theory and Adaptation Model The trainings prepared by the researcher in line with the literature information were held in 3 sessions. will be realized.Trainings are held in a classroom setting for 4 weeks and 2 lessons per session hour (100 minutes) in duration.

DETAILED DESCRIPTION:
The aim of the study was to teach nursing students nursing theories through creative drama method. The aim of the study was to investigate the effect of the teaching on the level of knowledge and perception of nursing profession. In the research A mixed research method using both quantitative and qualitative methods will be used.

The quantitative dimension of the research is a randomized controlled experimental study (pretest-posttest control group design). The qualitative dimension will consist of individual interviews with the experimental and control groups.

Hypotheses of the Study H1A: Teaching nursing theories with creative drama method increases the knowledge level of the students compared to the traditional method.

H1B: Teaching nursing theories with creative drama method compared to the traditional method increases students' perception of profession scores.

H1A0: Creative drama method compared to traditional method in teaching nursing theories has no effect on students' knowledge level scores.

H1B0: Creative drama method compared to traditional method in teaching nursing theories There is no effect of teaching with the use of the "vocational perception" method on students' vocational perception scores.

Haliç University Faculty of Health Sciences Nursing It will be conducted with the 1st year students of the Turkish Department between February and May 2024. The research population will be Haliç University Health Sciences in the 2023-2024 academic year.

First-year undergraduate students studying at the Faculty of Nursing, Department of Nursing (n=90). 25 people who meet the criteria, considering that there may be absenteeism during the data collection process.

It is planned to be conducted with a total of 50 students, 25 experimental and 25 control.

ELIGIBILITY:
Inclusion Criteria:

* Being a 1st year nursing student in Turkish Speak and understand Turkish Willingness to be involved in the study

Exclusion Criteria:

* To be a graduate of health vocational high school nursing and other health professions Having creative drama education Having a nursing model / theory education Having a psychological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Nursing Profession Perception Scale | 15 minutes
  "Nursing Profession Perception Scale" It is a 5-point Likert-type scale and consists of 22 items and two subscales; "Professional Qualifications and Professional Status". The "Professional Qualifications" subscale consists of items 1, 2, 3, 4, 5, 9, 10, 11, 13, 14, 15, 16, 17, 18, 19, 20, 21, and the "Professional Status" subscale consists of items 6, 7, 8, 12, 22. The statements used to determine the degree of perception The scoring is as follows: 1. Strongly disagree (1 point), 2. Disagree (2 points), 3.
  Undecided (3 points), 4. Agree (4 points), 5. Strongly Agree (5 points). The most The highest score was 110, the lowest score was 22, and the highest score of the "Professional Qualifications" sub-dimension (17 items) was 110. The highest score of the "Professional Status" sub-dimension (5 items) was 85 and the lowest score was 17. score is 25 and the lowest score is 5. The higher the total score obtained from the scale, the higher the occupational perception is positive.
The survey consists of 20 multiple-choice questions. | 30 minutes
  In line with the knowledge of the literature, the researcher has determined that nursing students to measure the level of knowledge before and after the training about the model / theories The survey consists of 20 multiple-choice questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Sevinç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevinc E, Ilhan SE. The effect of creative drama-based teaching on the knowledge level of nursing theories and perception of the nursing profession in a basic nursing course: A randomised controlled trial. Nurse Educ Pract. 2025 Dec 23;91:104679. doi: 10.1016/j.nepr.2025.104679. Online ahead of print. PMID 41455363